CLINICAL TRIAL: NCT05620836
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Efficacy and Safety Study of Povorcitinib (INCB054707) in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Efficacy and Safety of Povorcitinib (INCB054707) in Participants With Moderate to Severe Hidradenitis Suppurativa (HS)
Acronym: STOP-HS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 54707-302; 2022-501753-36-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; HS; INCB054707; Povorcitinib; Acne inversa; Hidradenitis
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 to Povorcitinib Dose A, Povorcitinib Dose B, or Placebo once a day (QD); participants who complete the placebo-controlled (PC) 12-week period may continue to a 42-week extension (EXT) period with Povorcitinib (Dose A or Dose B) QD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Povorcitinib Dose A (Experimental): Participants will receive Povorcitinib Dose A for 54 weeks.
  Interventions: Drug: Povorcitinib
- Povorcitinib Dose B (Experimental): Participants will receive Povorcitinib Dose B for 54 weeks.
  Interventions: Drug: Povorcitinib
- Placebo (Placebo Comparator): Participants will receive Placebo for 12 weeks, followed by Povorcitinib (Dose A or Dose B) for 42 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Povorcitinib — Oral, Tablet
  Other Names: INCB054707
  Arms: Povorcitinib Dose A; Povorcitinib Dose B
Drug: Placebo — Oral, Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Povorcitinib (INCB054707) in participants with moderate to severe Hidradenitis Suppurativa (HS) over a 12-week placebo-controlled period, followed by a 42-week extension period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years of age.
* Diagnosis of moderate to severe HS ≥ 3 months prior to Screening visit.
* HS lesions present in ≥ 2 distinct anatomic areas, 1 of which must be at least Hurley Stage II or Hurley Stage III, at both the Screening and Baseline visits.
* Total abscess and inflammatory nodule (AN) count ≥ 5 at both the Screening and Baseline visits.
* History of inadequate response to an appropriate course of at least 1 conventional systemic therapy for HS (or demonstrated intolerance to, or have a contraindication to, a conventional systemic therapy for HS)
* Agree to not use certain topical antiseptics on the areas affected by HS lesions during the placebo-controlled period.
* Willingness to avoid pregnancy or fathering children.
* Other inclusion criteria apply.

Exclusion Criteria:

* Draining tunnel count of > 20 at Screening or Baseline visits.
* Women who are pregnant (or who are considering pregnancy) or breastfeeding.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction; venous and arterial thrombosis, deep vein thrombosis, pulmonary embolism, stroke, moderate to severe heart failure, cerebrovascular accident, myocardial infarction, or other significant cardiovascular diseases; Q-wave interval abnormalities; disseminated herpes zoster or dermatomal herpes zoster; disseminated herpes simplex; chronic/recurrent infections; malignancies.
* Evidence of infection with TB, HBV, HCV or HIV.
* History of failure to JAK inhibitor treatment of any inflammatory disease.
* Laboratory values outside of the protocol-defined ranges.
* Other exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response (HiSCR) | Week 12
  HiSCR is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.

SECONDARY OUTCOMES:
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | Week 12
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Proportion of participants with flare | 12 Weeks
  Participants who experience at least 1 flare over 12 weeks; flare is defined as at least a 25% increase in the total abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline.
Proportion of participants with a ≥ 3-point decrease in Skin Pain Numeric Rating Scale (NRS) score among participants with baseline Skin Pain NRS score ≥ 3 | Week 12
  Participants with a Skin Pain score of at least 3 at baseline and who experience at least a 3-point decrease in Skin Pain score at Week 12, relative to baseline. Skin Pain is an 11-point NRS, ranging from 0 (no skin pain) to 10 (worst skin pain).
Proportion of participants who achieve Skin Pain NRS30 at Week 12 among participants with baseline Skin Pain NRS score ≥ 3. | Week 12
  Participants with a Skin Pain score of at least 3 at baseline and who achieve at Week 12 Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Proportion of participants with a ≥ 4-point increase from baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score | Week 12
  Participants with a baseline FACIT-F score ≤ 48 and who experience at least a 4-point increase in FACIT-F score at Week 12, relative to baseline. The FACIT-F scale is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days, with scores ranging from 0 (worst fatigue) to 52 (no fatigue).
Mean change from baseline in Dermatology Life Quality Index (DLQI) score | 54 weeks
  The DLQI is a skin disease specific questionnaire aimed at the evaluation of how symptoms and treatment affect participants' health-related quality of life (QoL). The DLQI total score ranges from 0 to 30, with higher scores indicating lower skin health related QoL.
Mean change from baseline in abscess count | 54 weeks
  Defined as mean change of abscess(es) count relative to baseline.
Percentage change from baseline in abscess count | 54 weeks
  Percent Change from baseline in number of abscess(es)
Mean change from baseline in inflammatory nodule count | 54 weeks
  Defined as mean change of inflammatory nodule count relative to baseline.
Percentage change from baseline in inflammatory nodule count | 54 weeks
  Defined as percent change from baseline in number of inflammatory nodule(s)
Mean change from baseline in draining tunnel count | 54 weeks
  Defined as mean change of draining tunnel count relative to baseline.
Percentage change from baseline in draining tunnel count | 54 weeks
  Defined as Percent change from baseline in number of draining tunnel(s)
Extension Period: Proportion of participants who achieve HiSCR | Week 24
  HiSCR is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants who achieve HiSCR75 | Week 24
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants with flare | From Week 12 through Week 24
  Participants who experience at least 1 flare over the period under assessment; flare is defined as at least a 25% increase in the total abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline.
Extension Period: Proportion of participants who achieved Skin Pain NRS30 among participants with baseline Skin Pain NRS score ≥ 3. | Week 24
  Skin Pain NRS30 defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Extension Period: Proportion of participants who achieve HiSCR | Week 54
  HiSCR is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants who achieve HiSCR75 | Week 54
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants with flare | From Week 12 through Week 54
  Participants who experience at least 1 flare over the period under assessment; flare is defined as at least a 25% increase in the total abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline
Extension Period: Proportion of participants who achieved Skin Pain NRS30 among participants with baseline Skin Pain NRS score ≥ 3. | Week 54
  Participants with a Skin Pain score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Extension Period: Proportion of participants who achieve maintenance of HiSCR or greater response at each visit | From Week 12 through Week 54
  Maintenance of response defined as participants who achieve HiSCR at Week 12 and maintain it or achieve greater response at each visit during the EXT period.
Extension Period: Proportion of participants who achieve maintenance of HiSCR75 or greater response at each visit | From Week 12 through Week 54
  Maintenance of response defined as participants who achieve HiSCR75 at Week 12 and maintain it or achieve greater response at each visit during the EXT period.

CONTACTS AND LOCATIONS:
Locations (101):
- United States (38):
  - Investigative Site US240, Scottsdale, Arizona
  - Investigative Site US237, Scottsdale, Arizona
  - Investigative Site US214, Arkansas City, Arkansas
  - Investigative Site US242, Fayetteville, Arkansas
  - Investigative Site US223, Los Angeles, California
  - Investigative Site US226, San Diego, California
  - Investigative Site US222, San Francisco, California
  - Investigative Site US233, Washington D.C., District of Columbia
  - Investigative Site US228, Brandon, Florida
  - Investigative Site US227, Margate, Florida
  - Investigative Site US204, Miami, Florida
  - Investigative Site US236, Miami, Florida
  - Investigative Site US200, Ocala, Florida
  - Investigative Site US201, Tampa, Florida
  - Investigative Site US220, West Dundee, Illinois
  - Investigative Site US206, Indianapolis, Indiana
  - Investigative Site US241, Iowa City, Iowa
  - Investigative Site US209, Louisville, Kentucky
  - Investigative Site US207, Metairie, Louisiana
  - Investigative Site US229, New Orleans, Louisiana
  - Investigative Site US224, Baltimore, Maryland
  - Investigative Site US208, Beverly, Massachusetts
  - Investigative Site US221, Quincy, Massachusetts
  - Investigative Site US213, Detroit, Michigan
  - Investigative Site US217, Waterford, Michigan
  - Investigative Site US212, Minneapolis, Minnesota
  - Investigative Site US239, Omaha, Nebraska
  - Investigative Site US230, Hightstown, New Jersey
  - Investigative Site US202, New York, New York
  - Investigative Site US210, Rochester, New York
  - Investigative Site US205, Chapel Hill, North Carolina
  - Investigative Site US215, Bexley, Ohio
  - Investigative Site US203, Columbus, Ohio
  - Investigative Site US232, Murfreesboro, Tennessee
  - Investigative Site US235, Arlington, Texas
  - Investigative Site US218, Bellaire, Texas
  - Investigative Site US238, Pflugerville, Texas
  - Investigative Site US234, San Antonio, Texas
- Australia (8):
  - Investigative Site AU205, Kogarah, New South Wales
  - Investigative Site AU203, Kotara, New South Wales
  - Investigative Site AU200, Liverpool, New South Wales
  - Investigative Site AU202, Benowa, Queensland
  - Investigative Site AU206, Woolloongabba, Queensland
  - Investigative Site AU207, Woolloongabba, Queensland
  - Investigative Site AU201, Carlton, Victoria
  - Investigative Site AU204, Melbourne, Victoria
- Bulgaria (5):
  - Investigative Site BG203, Sofia
  - Investigative Site BG202, Sofia
  - Investigative Site BG200, Sofia
  - Investigative Site BG204, Sofia
  - Investigative Site BG201, Stara Zagora
- Canada (8):
  - Investigative Site CA202, Calgary, Alberta
  - Investigative Site CA204, Edmonton, Alberta
  - Investigative Site CA200, Surrey, British Columbia
  - Investigative Site CA205, Fredericton, New Brunswick
  - Investigative Site CA207, Mississauga, Ontario
  - Investigative Site CA208, Richmond Hill, Ontario
  - Investigative Site CA206, Saint-Jérôme, Quebec
  - Investigative Site CA203, St. John's
- Denmark (2):
  - Investigative Site DK200, Århus N
  - Investigative Site DK201, Roskilde
- France (7):
  - Investigative Site FR200, Antony
  - Investigative Site FR205, Dijon
  - Investigative Site FR204, Lyon
  - Investigative Site FR203, Nice
  - Investigative Site FR206, Reims
  - Investigative Site FR202, Rouen
  - Investigative Site FR201, Toulon
- Germany (10):
  - Investigative Site US225, Frankfurt am Main, MA
  - Investigative Site DE202, Berlin
  - Investigative Site DE203, Bochum
  - Investigative Site DE201, Dessau
  - Investigative Site DE207, Erlangen
  - Investigative Site DE208, Göttingen
  - Investigative Site DE205, Heidelberg
  - Investigative Site DE200, Kiel
  - Investigative Site DE204, Lübeck
  - Investigative Site DE206, Mainz
- Italy (8):
  - Investigative Site IT200, Ancona
  - Investigative Site IT204, Brescia
  - Investigative Site IT207, Catania
  - Investigative Site IT202, Milan
  - Investigative Site IT203, Napoli
  - Investigative Site IT206, Pisa
  - Investigative Site IT205, Roma
  - Investigative Site IT201, Rozzano
- Poland (4):
  - Investigative Site PL203, Lublin
  - Investigative Site PL200, Rzeszów
  - Investigative Site PL201, Warsaw
  - Investigative Site PL202, Warsaw
- Spain (6):
  - Investigative Site ES203, Alicante
  - Investigative Site ES202, Las Palmas de Gran Canaria
  - Investigative Site ES204, Madrid
  - Investigative Site ES201, Madrid
  - Investigative Site ES205, Madrid
  - Investigative Site ES200, Manises
- United Kingdom (5):
  - Investigative Site GB202, Birmingham
  - Investigative Site GB200, Dudley
  - Investigative Site GB201, Leeds
  - Investigative Site GB204, London
  - Investigative Site GB203, Salford

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Efficacy and Safety of Povorcitinib (INCB054707) in Participants With Moderate to Severe Hidradenitis Suppurativa (HS) — https://incyteclinicaltrials.com/studies/incb-54707-302